CLINICAL TRIAL: NCT03016715
Title: A Prospective, Double-Blind, Cross-Over, Pilot Study to Assess Safety and Efficacy of Topical Sirolimus 2% in the Treatment of Plantar Blistering in Patients With Epidermolysis Bullous Simplex (EBS)
Brief Title: Using Topical Sirolimus 2% for Patients With Epidermolysis Bullous Simplex (EBS) Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Premier Specialists, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-05-413
Record Dates: First submitted 2017-01-09; First posted 2017-01-10 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Epidermolysis Bullosa Simplex; Epidermolysis Bullosa Simplex Kobner; Weber-Cockayne Syndrome
Keywords: Epidermolysis bullosa simplex
MeSH Terms: conditions — Epidermolysis Bullosa Simplex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Sirolimus, 2% topical ointment will be used during randomization
  Interventions: Drug: Sirolimus 2%
- Vehicle (Placebo Comparator): A placebo topical ointment will be used during randomization.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Sirolimus 2%
  Arms: Treatment
Drug: Vehicle
  Other Names: Placebo
  Arms: Vehicle

SUMMARY:
: Epidermolysis bullosa (EB) simplex is a rare orphan disease caused by a mutation in DNA leading to abnormal dominant keratins in the skin. Patients with EB simplex develop lifelong painful thick soles on their feet, and current standard of care is supportive. This pilot study will target the dominant mutant keratin proteins in the skin to ameliorate the severity of EB simplex. The purpose is to improve the function of EB simplex feet with an application of topical sirolimus, 2%. The investigators plan on inhibiting the mTOR pathway to down regulate the translation of defective keratin proteins and work through anti proliferative pathways.

DETAILED DESCRIPTION:
The proposed 40 week pilot study being conducted is a prospective, double-blind, randomized, placebo-controlled crossover study. Participants will be assigned to treat both feet with either topical sirolimus, 2% cream daily or placebo (vehicle-control) for 12 weeks, followed by a 4 week washout period, then re-treatment to both feet will occur by the cross-over intervention.

These studies will exploit the naturally occurring transcriptional regulation of keratin sequences, the known gene aberration causing EB simplex, and assess the potential for mTOR pathway inhibition in treatment of the patient's plantar lesions. The objective of this study is to assess (1) the safety of topical rapamycin for plantar lesions for the treatment of EB simplex, and 2) test if topical rapamycin to improves the clinical severity of lesional skin, including pain and itch, in subjects with EB simplex at the end of treatment versus baseline and compared to an intrasubject placebo treated control. Wound size measurement, quality of life evaluation will be assessed using epidermolysis bullosa (QOLEB), and EB disease activity and Scarring Index (EBDASI). With the results of this pilot study, physicians would be able to transition from supportive care (the current state of the art for EB simplex) to targeted molecular therapeutics, leading to improved mobility and quality of life for patients with EB simplex.

ELIGIBILITY:
Inclusion Criteria:

Subjects must:

* Be capable of understanding the purpose and risks of the study and sign a written Informed Consent Form (ICF); Legally authorized representative of subjects willing and able to give consent for children 5-18 yo
* Be male or female with a diagnosis of EBS
* Minimum EBDASI feet activity score of 2/10
* Age - 5 years or older
* Ability to complete 12 study visits within a 40-week period, each for approximately 30-60 minutes.

Anticipated life expectancy ≥52 weeks

* Males and females of childbearing potential should be using an effective means of contraception.
* Laboratory values within the range of normal for the participating institution unless the PI feels they are not clinically relevant
* Be able to comply with all study requirements

Exclusion Criteria:

* Allergy to sirolimus or components of the vehicle ointment
* Pregnancy, breast feeding
* Prior history of liver disease
* Serious known concurrent medical illness or infection, which could potentially present a safety risk and/or prevent compliance with the requirements of the treatment program.
* Known immunodeficiency virus or syndrome including those with:
* Acquired Immunodeficiency Syndrome (AIDS)
* Human Immunodeficiency Virus (HIV)
* Hepatitis B
* Prior history of grafting surgeries or other surgeries in the dermatologic treatment area
* History of significant condition in the dermatologic treatment area such as trauma, which could impair evaluation for the treatment of EBS or non-healing chronic wound.
* Use of other investigational drugs within 30 days of the screening visit and/or has not recovered from any side effects of prior investigational drugs or procedure in the affected area (e.g., a biopsy).
* Use of acitretin within the last 1 month
* Use of Roaccutane within last 3 months
* Botox injections to the feet within the last 6 months.
* Participant is planning extra physical activities within the next 3 months.
* Amputated foot

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Foot Health Status Questionnaire | Change from Baseline to End of Treatment completion at 32 Week
  Foot function utilizing the validated Foot Health Status Questionnaire (FHSQ) as a change from baseline to the end of each treatment.

SECONDARY OUTCOMES:
FitBit® / pedometer | Baseline and through study treatment completion at 32-weeks]
Plantar defect size using 3D Photography | Change in total defect area from Baseline, clinical visits at Week 4, Week 12, Week 16, Week 28, through study treatment completion at 32-weeks
  Plantar defect size measurements using 3D photography (% change in total defect area) from baseline to the end of each treatment.
Child Dermatological Quality of Life Questionnaire | Baseline through study treatment completion at 32 weeks
The Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI) Disease Severity Scale | Baseline and through study treatment completion at 32-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dedee F Murrell, MD, Study Chair — University of New South Wales
Locations (1):
- Premier Specialists, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Fine JD, Bruckner-Tuderman L, Eady RA, Bauer EA, Bauer JW, Has C, Heagerty A, Hintner H, Hovnanian A, Jonkman MF, Leigh I, Marinkovich MP, Martinez AE, McGrath JA, Mellerio JE, Moss C, Murrell DF, Shimizu H, Uitto J, Woodley D, Zambruno G. Inherited epidermolysis bullosa: updated recommendations on diagnosis and classification. J Am Acad Dermatol. 2014 Jun;70(6):1103-26. doi: 10.1016/j.jaad.2014.01.903. Epub 2014 Mar 29. PMID 24690439
- [Background] Fine JD, Johnson LB, Weiner M, Suchindran C. Assessment of mobility, activities and pain in different subtypes of epidermolysis bullosa. Clin Exp Dermatol. 2004 Mar;29(2):122-7. doi: 10.1111/j.1365-2230.2004.01428.x. PMID 14987264
- [Background] Lane EB, McLean WH. Keratins and skin disorders. J Pathol. 2004 Nov;204(4):355-66. doi: 10.1002/path.1643. PMID 15495218
- [Background] Castedo M, Ferri KF, Kroemer G. Mammalian target of rapamycin (mTOR): pro- and anti-apoptotic. Cell Death Differ. 2002 Feb;9(2):99-100. doi: 10.1038/sj.cdd.4400978. No abstract available. PMID 11840159
- [Background] Guba M, von Breitenbuch P, Steinbauer M, Koehl G, Flegel S, Hornung M, Bruns CJ, Zuelke C, Farkas S, Anthuber M, Jauch KW, Geissler EK. Rapamycin inhibits primary and metastatic tumor growth by antiangiogenesis: involvement of vascular endothelial growth factor. Nat Med. 2002 Feb;8(2):128-35. doi: 10.1038/nm0202-128. PMID 11821896
- [Background] Fogel AL, Hill S, Teng JM. Advances in the therapeutic use of mammalian target of rapamycin (mTOR) inhibitors in dermatology. J Am Acad Dermatol. 2015 May;72(5):879-89. doi: 10.1016/j.jaad.2015.01.014. Epub 2015 Mar 11. PMID 25769191
- [Background] Raught B, Gingras AC, Sonenberg N. The target of rapamycin (TOR) proteins. Proc Natl Acad Sci U S A. 2001 Jun 19;98(13):7037-44. doi: 10.1073/pnas.121145898. PMID 11416184
- [Background] Hickerson RP, Leake D, Pho LN, Leachman SA, Kaspar RL. Rapamycin selectively inhibits expression of an inducible keratin (K6a) in human keratinocytes and improves symptoms in pachyonychia congenita patients. J Dermatol Sci. 2009 Nov;56(2):82-8. doi: 10.1016/j.jdermsci.2009.07.008. Epub 2009 Aug 21. PMID 19699613
- [Background] Riskowski JL, Hagedorn TJ, Hannan MT. Measures of foot function, foot health, and foot pain: American Academy of Orthopedic Surgeons Lower Limb Outcomes Assessment: Foot and Ankle Module (AAOS-FAM), Bristol Foot Score (BFS), Revised Foot Function Index (FFI-R), Foot Health Status Questionnaire (FHSQ), Manchester Foot Pain and Disability Index (MFPDI), Podiatric Health Questionnaire (PHQ), and Rowan Foot Pain Assessment (ROFPAQ). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S229-39. doi: 10.1002/acr.20554. No abstract available. PMID 22588747
- [Background] Loh CC, Kim J, Su JC, Daniel BS, Venugopal SS, Rhodes LM, Intong LR, Law MG, Murrell DF. Development, reliability, and validity of a novel Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI). J Am Acad Dermatol. 2014 Jan;70(1):89-97.e1-13. doi: 10.1016/j.jaad.2013.09.041. PMID 24355263
- [Background] Venugopal SS, Yan W, Frew JW, Cohn HI, Rhodes LM, Tran K, Melbourne W, Nelson JA, Sturm M, Fogarty J, Marinkovich MP, Igawa S, Ishida-Yamamoto A, Murrell DF. A phase II randomized vehicle-controlled trial of intradermal allogeneic fibroblasts for recessive dystrophic epidermolysis bullosa. J Am Acad Dermatol. 2013 Dec;69(6):898-908.e7. doi: 10.1016/j.jaad.2013.08.014. Epub 2013 Sep 24. PMID 24075228
- [Background] Frew JW, Martin LK, Nijsten T, Murrell DF. Quality of life evaluation in epidermolysis bullosa (EB) through the development of the QOLEB questionnaire: an EB-specific quality of life instrument. Br J Dermatol. 2009 Dec;161(6):1323-30. doi: 10.1111/j.1365-2133.2009.09347.x. Epub 2009 Jun 11. PMID 19681875
- [Background] Elman S, Hynan LS, Gabriel V, Mayo MJ. The 5-D itch scale: a new measure of pruritus. Br J Dermatol. 2010 Mar;162(3):587-93. doi: 10.1111/j.1365-2133.2009.09586.x. Epub 2009 Dec 1. PMID 19995367
- [Background] Storm FA, Heller BW, Mazza C. Step detection and activity recognition accuracy of seven physical activity monitors. PLoS One. 2015 Mar 19;10(3):e0118723. doi: 10.1371/journal.pone.0118723. eCollection 2015. PMID 25789630